CLINICAL TRIAL: NCT05966727
Title: Exploratory Evaluation of the Effect of Cholestyramine on Serum Levels of Persistent Organic Pollutants in Obese Female Patients - OBESE (OBesity, CholEStyramine, WomEn)
Brief Title: Exploratory Evaluation of the Effect of Cholestyramine on Serum Levels of POPs in Obese Female Patients
Acronym: OBESE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-AOI-07
Record Dates: First submitted 2023-07-05; First posted 2023-08-01 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Abdominal; Diabetes; Bariatric Surgery Candidate
Keywords: endocrine disrupter; Obesity; Diabetes; Bariatric Surgery
MeSH Terms: conditions — Obesity, Abdominal; Diabetes Mellitus; Obesity | interventions — Cholestyramine Resin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cholestyramine intake (Experimental): 1 sachet (4 grams) 3 times a day, corresponding to a daily dose of 12 grams. Preferably taken at mealtimes.
  Treatment lasts 4 months.
  Interventions: Drug: Cholestyramine Powder

INTERVENTIONS:
Drug: Cholestyramine Powder — Bile salt chelating resin, used as a lipid-lowering treatment.
  Other Names: Questran

SUMMARY:
Environmental endocrine disruptors (EDCs) represent a major problem for human health.Some PEEs can accumulate in the fatty tissue of the human body thanks to their lipophilic nature, and are known as persistent organic pollutants (POPs).

To assess the benefit of cholestyramine treatment on POPs blood levels in obese patients of childbearing age undergoing bariatric surgery, in order to reduce their preoperative POPs load more rapidly. Indeed, the investigators hypothesize that cholestyramine is capable, outside of acute exposure accidents, of promoting the elimination and release of POPs in the human population. Given this hypothesis, a treatment administered prior to bariatric surgery could reduce pre-operative plasma levels of POPs and thus, in fine, minimize the concentrations reached post-operatively, which are dependent on the release induced by lipolysis (massive and rapid weight loss) and pre-operative plasma concentrations.

DETAILED DESCRIPTION:
Environmental endocrine disruptors (EDCs) represent a major problem for human health. These chemical compounds from industry (pesticides, paints, plastics, etc.) are present in our daily lives, with exposure as early as foetal life. PEEs are capable of interfering with the endocrine system, but also of disrupting the signalling pathways of carbohydrate and lipid metabolism, and consequently of causing adverse effects on the health of an individual and/or his or her offspring. They are implicated in numerous pathologies, notably those linked to nervous system development, reproduction and chronic diseases such as obesity and diabetes. Thanks to their lipophilic nature, some PEEs can accumulate in the adipose tissue of the human body, and are known as persistent organic pollutants (POPs). Numerous longitudinal epidemiological studies have demonstrated higher concentrations of PEEs, particularly POPs, in obese and/or type 2 diabetic patients. In addition, these POPs pass easily across the placenta into fetal blood and, more readily, into breast milk. The developing fetus and infant are particularly sensitive to POPs, due to their lower volume of distribution and immature metabolism pathways.

In a recently published longitudinal study (PHRC POLOB), the investigators showed that massive weight loss during the first year after bariatric surgery is associated with a prolonged release of POPs from adipose tissue, directly dependent on pre-operative plasma levels. For some compounds, this release exceeds the health reference values set by ANSES, even one year after surgery. Short- and long-term consequences must therefore be considered, particularly for obese women of childbearing age (60% of the population undergoing bariatric surgery), because of the risks to the health of the unborn child in the event of pregnancy occurring early after surgery, even if a 6-month delay is recommended between surgery and the planning of a pregnancy.

While health education is an important lever for limiting daily exposure, identifying a treatment that can reduce the degree of exposure to EEPs is crucial, especially in a population where pregnancy is planned in the short term. Cholestyramine is a bile salt chelating resin used as a lipid-lowering treatment. It has been used off-label in a case of accidental acute contamination by certain POPs, reducing plasma levels without adverse effects, by promoting elimination through interaction with the enterohepatic cycle.

The investigators hypothesize that cholestyramine is capable, outside of acute exposure events, of promoting the elimination and release of POPs in the human population. Given this hypothesis, a treatment administered prior to bariatric surgery could reduce pre-operative plasma levels of POPs and thus, ultimately, minimize the concentrations reached post-operatively, which are dependent on lipolysis-induced release (massive and rapid weight loss) and pre-operative plasma concentrations. To confirm this hypothesis, the investigators propose to evaluate in an exploratory way, on a selected cohort of patients, the effect of pre-operative cholestyramine treatment on serum concentrations of different POPs before and after bariatric surgery.

If the results of this proof-of-concept study are positive, it will be possible to pursue the study of cholestyramine with more powerful and comparative studies, with a view to eventually considering a treatment to reduce the potentially harmful risks of POPs in cases of confirmed pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with a retained indication for bariatric surgery (BMI > 40 kg/m2 or BMI > 35 kg/m2 with complication(s) amenable to improvement by surgery)
* Aged between 18 and 45
* Using effective contraception (oral contraception, hormonal or non-hormonal intrauterine device, progestin implant), which will be adapted in the perioperative period in accordance with current recommendations (HAS, BARIA-MAT)
* Affiliated to a social security scheme
* Have signed an informed consent form

Exclusion Criteria:

* Pregnant (urine pregnancy test) or breast-feeding women
* Known allergy or intolerance to cholestyramine
* Chronic constipation
* Chronic pathology likely to interfere with treatment efficacy (unbalanced diabetes characterized by HbA1c > 7%, known and treated dyslipidemia, chronic renal insufficiency with GFR < 60 ml/min, hepatocellular insufficiency)
* Patients receiving anti-vitamin K, digoxin or levothyroxine therapy, or likely to receive such therapy within 3 months of inclusion.
* Phenylketonuria
* Inability to give consent
* Patient under legal protection (guardianship, curatorship, safeguard of justice...)
* Patient deprived of liberty by judicial or administrative decision,
* Patients under psychiatric care which makes it impossible for them to consent to participation, or who are hospitalized under duress.
* Participation in another interventional study (outside the PaCO project).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Measurement of serum persistent organic pollutants (POPs) concentrations by mass spectrometry. | 19 month
  Evaluation of the effect of cholestyramine treatment on serum concentrations of various persistent organic pollutants (POPs) in a population of population of obese women of childbearing age for whom bariatric surgery is bariatric surgery is indicated.

SECONDARY OUTCOMES:
Measurement of serum POPs concentrations by mass spectrometry after bariatric surgery | 19 month
  Evaluation of the effect of pre-operative cholestyramine treatment with respect to observed and expected post-bariatric surgery salting-out.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas CHEVALIER, Principal Investigator — CHU NICE
Locations (1):
- CHU Nice - Hôpital de l'Archet 2, Nice, Alpes-Mritimes, France